CLINICAL TRIAL: NCT02936817
Title: A Study to Assess the Effect of the Aerobika® Device in Addition to Standard of Care Treatment in Sputum Producing COPD Patients Using Functional Respiratory Imaging (FRI)
Brief Title: Study to Assess the Effect of the Aerobika Device in Addition to Standard of Care Treatment in Sputum Producing COPD Patients Using FRI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: FLUIDDA nv (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLUI-2016-166
Record Dates: First submitted 2016-10-13; First posted 2016-10-18 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive; COPD
Keywords: HRCT; High Resolution Computed Tomography scans; Functional Respiratory Imaging; CT scan; Computed Tomography; COPD; sputum producing COPD patients; Aerobika® device
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aerobika® device (Other): For a period of 15 +/- 3 days all subjects will use the Aerobika® device before administration of their stable standard of care treatment regimen (i.e. study patients should use the device before each inhalation medication administration, with a minimum use of the device of twice daily). HRCT scans wil be taken at visit 1 and visit 3.
  Interventions: Device: Aerobika® Device; Radiation: HRCT scans

INTERVENTIONS:
Device: Aerobika® Device — For a period of 15 +/- 3 days subjects will use the Aerobika® device before administration of their stable standard of care treatment regimen (i.e. study patients should use the device before each inhalation medication administration, with a minimum use of the device of twice daily).
  Other Names: Aerobika® Oscillating Positive Expiratory Pressure Therapy System
Radiation: HRCT scans — A HRCT scan at Functional Residual Capacity (FRC) and Total Lung Capacity (TLC) will be taken on visit 1, and visit 3. An upper airway (UA) scan will be taken on visit 1.
  Other Names: High Resolution Computed Tomography scans

SUMMARY:
Primary:

The primary objective of this study is to evaluate the effect of the Aerobika® device on the aerosol deposition pattern of concomitant inhalation medication using FRI.

Secondary:

The secondary objective of this study is to evaluate the effect of the Aerobika® device on the airway volume (iVaw), lung and lobe volume (iVlobes), airway resistance (iRaw), hyperinflation, airway wall thickness (iVaww), blood vessel density (iVbv), and air trapping using FRI.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject ≥ 40 and ≤ 85 years old.
2. Written informed consent obtained.
3. Subject with a documented diagnosis of COPD with GOLD II to IV severity according to the GOLD guidelines,
4. Subject with a cooperative attitude and ability to be trained to correctly use the Aerobika® device.
5. Female subject t of childbearing potential must confirm that a contraception method was used at least 14 days before Visit 1 and will continue to use a contraception method during the study.
6. Subject must be sputum producing and treated in accordance with the GOLD guidelines. Sputum producing subjects are defined as patients who report productive cough with sputum "several days a week" (>2 days a week) or "almost every day" in the month prior to the study.
7. Subject must be able to understand and complete the protocol requirements, instructions and protocol-stated restrictions.
8. Subject must use standard of care treatment. The regime of standard of care treatment must be on a stable dose of medication at least 1 week before Visit 1.
9. Subject should have unchanged smoking status within 3 months of Visit 1 and throughout the study period.

Exclusion Criteria:

1. Pregnant or lactating female.
2. Subject with upper or lower airway infection that has not resolved within 4 weeks of the Screening Visit.
3. Subject experiencing an exacerbation defined as an acute change in the patient 's baseline dyspnea, cough, and/or sputum that is beyond normal day to day variations and necessitates the administration or doubling of systemic corticosteroid treatment within 4 weeks of the Screening Visit.
4. Subjects unable to tolerate the increased work of breathing.
5. Subject with a history of cerebrovascular disease
6. Patient with clinical significant hemodynamic instability (i.e. blood pressure instability).
7. Subject with recent facial, oral, or skull surgery or trauma.
8. Subject with active acute sinusitis.
9. Subject with active epistaxis (i.e. bleeding nose).
10. Subject with a history of esophageal surgery.
11. Subject with an active diagnosis of nausea on Visit 1.
12. Subject with active hemoptysis (i.e. bleeding from lungs).
13. Subject with untreated pneumothorax (i.e. untreated collapsed lung).
14. Subject with known or suspected tympanic membrane rupture or other middle ear pathology.
15. Subject unable to perform pulmonary function testing.
16. Subject with an uncontrolled disease or any condition that might, in the judgement of the investigator, place the patient at undue risk or potentially compromise the results or interpretation of the study.
17. Subject with active cancer or any other chronic disease with poor prognosis and /or affecting patient status
18. Subject unlikely to comply with the protocol or unable to understand the nature, scope, and possible consequences of the study.
19. Subject who received any investigational new drug within 4 weeks of Visit 1 or twice the duration of the biological effect of any drug (whichever is longer).
20. Subject with a history of alcohol or substance abuse that, in the opinion of the investigator, may be of clinical significance.
21. Subject who has undergone major surgery within 12 weeks of Visit 1 or has planned to undergo a major surgery before the end of the study.
22. Subject with diagnosis of asthma.
23. Inability to correctly use the sham device.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Changes in the number of deposited particles of concomitant inhalation medication per pre-defined airway section | At day 1 and after 15 +/- 3 days of treatment
  FRI parameters: HRCT scan will be taken at visit 1 and visit 3.

SECONDARY OUTCOMES:
Changes in Distal airway volumes (iVaw) | At day 1 and after 15 +/- 3 days of treatment
  FRI parameters: HRCT scan will be taken at visit 1 and visit 3.
Changes in Distal airway resistance (iRaw) | At visit 1 and after 15 +/- 3 days of treatment
  FRI parameters: HRCT scan will be taken at visit 1 and visit 3.
Changes in Lung and Lobe Volumes (iVlobes) | At day 1 and after 15 +/- 3 days of treatment
  FRI parameters: HRCT scan will be taken at visit 1 and visit 3.
Changes in Airway Wall Thickness (iVaww) | At day 1 and after 15 +/- 3 days of treatment
  FRI parameters: HRCT scan will be taken at visit 1 and visit 3.
Changes in Blood Vessel Density (iVbv) | At day 1 and after 15 +/- 3 days of treatment
  FRI parameters: HRCT scan will be taken at visit 1 and visit 3.
Changes in Air Trapping | At day 1 and after 15 +/- 3 days of treatment
  FRI parameters: HRCT scan will be taken at visit 1 and visit 3.
Changes in Forced Expiratory Volume in 1 Second (FEV1) | At day 1 and after 15 +/- 3 days of treatment
  Spirometry parameter
Changes in Forced Vital Capacity (FVC) | At day 1 and after 15 +/- 3 days of treatment
  Spirometry parameter
Changes in Peak Expiratory Flow (PEF) | At day 1 and after 15 +/- 3 days of treatment
  Spirometry parameter
Changes in Forced Expiratory Flow between 25% to 75% of FVC (FEF 25-75) | At day 1 and after 15 +/- 3 days of treatment
  Spirometry parameter
Changes in Inspiratory Capacity (IC) | At day 1 and after 15 +/- 3 days of treatment
  Spirometry parameter
Changes in Tiffeneau Index (FEV1/FVC ratio) | At day 1 and after 15 +/- 3 days of treatment
  Spirometry parameter
Changes in Functional Residual Capacity (FRC) | At day 1 and after 15 +/- 3 days of treatment
  Body plethysmography parameter
Changes in Total Lung Capacity (TLC) | At day 1 and after 15 +/- 3 days of treatment
  Body plethysmography parameter
Changes in Airway Resistance (Raw) | At day 1 and after 15 +/- 3 days of treatment
  Body plethysmography parameters: Airway resistance
Changes in Specific airway conductance (sGaw) | At day 1 and after 15 +/- 3 days of treatment
  Body plethysmography parameters: Airway resistance

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Backer, MD, PhD, Principal Investigator — University Hospital of Antwerp
Locations (1):
- University Hospital of Antwerp, Edegem, Antwerp, Belgium